CLINICAL TRIAL: NCT05084976
Title: Parental Perception of COVID-19 Vaccine in Pediatric Patients With Tracheostomy and Ventilator Dependence
Brief Title: Parental Perception of COVID-19 Vaccine in Technology Dependent Patients
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0822
Record Dates: First submitted 2021-10-18; First posted 2021-10-20 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Chronic Respiratory Failure; Tracheostomy Complication; Mechanical Ventilation Complication
Keywords: Technology dependent; Tracheostomy; Mechanical ventilator; Non invasive mechanical ventilator; Pediatric patient; COVID 19 vaccine; Vaccine hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric Technology Dependent Patients at Cohen Children's Medical Center
  Interventions: Behavioral: COVID 19 vaccine counseling
- Pediatric Technology Dependent Patients at Ann & Robert H. Lurie Children's Hospital of Chicago
  Interventions: Behavioral: COVID 19 vaccine counseling

INTERVENTIONS:
Behavioral: COVID 19 vaccine counseling — After surveys are completed, pulmonary provider (nurse practitioner or physician) will provide counseling via phone or in person about the COVID 19 vaccine. Safety, efficacy and side effects will be reviewed.

SUMMARY:
This study involves conducting a telephonic or in person survey regarding parental perception and attitudes about vaccinating the respective "technology dependent" child with the COVID 19 vaccination. "Technology dependent" includes tracheostomy dependence, artificial ventilator dependence and non invasive mechanical ventilation dependence. This population is vulnerable since most patients have underlying lung disease, chronic respiratory failure and require respiratory equipment to assist with breathing. "Technology dependent" patients are particularly vulnerable to respiratory infections and are considered high risk for developing severe COVID 19 illness. Despite this population's high risk for morbidity and mortality from respiratory viral infections, the investigator hypothesize that 50% of the parents are still vaccine hesitant.

DETAILED DESCRIPTION:
Vaccinating the population is the next step in combating COVID 19 pandemic however there continues to be vaccine hesitancy. Vaccine hesitancy is the indecision of consenting to vaccination (Dosanjh, 2021) and is not a new phenomenon. The most recent example is the reemergence of measles in the United States prior to the COVID 19 pandemic. Anti-vaccine groups have spread messages of conspiracy theories, myths and misperceptions, questions about the speed of vaccine development and long term side effects in the media which also attributes to COVID-19 vaccine hesitancy (Khubcandani et al, 2021).

Children infected with COVID 19 typically have mild symptoms of the disease. Risk factors associated with severe disease are neonatal age group, male gender, lower respiratory tract disease and pre-existing medical conditions. Children who use chronic home mechanical ventilation are considered a high-risk group for developing severe COVID 19 infection (Vasconcello-Castillo et al., 2020). These children have various diagnoses and pathologies such as neuromuscular disease, sleep disorders and chronic lung disease. These patients require continuous use of ventilatory support in the home and are at high risk for respiratory infections and mortality. Most of these patients need advanced nursing care and special respiratory equipment to prevent hospitalization such as manual chest physiotherapy, mechanical ex-sufflator device, chest vest device and increased ventilator support.

Recently the FDA approved of Pfizer's COVID 19 vaccine in ages 12 and older. It is anticipated that by fall 2021 the Pfizer COVID 19 vaccine will be approved by the FDA for children ages 2 and older. Vaccinating children will help decrease transmission of COVID 19, contribute to community immunity and allow kids go back to camps this summer and back to in-person school more safely.

Since the chronic home mechanical ventilation population is at risk for developing severe COVID 19 disease, the investigator would hypothesize that most parents are ready and willing to vaccinate their children. The purpose of this study is to evaluate the parental perception of COVID 19 vaccine in pediatric patients with "technology dependence" and identify the barriers to vaccination.

After surveys are collected and barriers are identified, vaccine counseling will be provided by a provider (nurse practitioner or physician). Vaccine safety, efficacy, side effects will be reviewed with the parents.

ELIGIBILITY:
Inclusion Criteria:

* Mother or father of child will be interviewed
* Pediatric patient (age 0-21)
* "Technology dependent" with one or more of the following: tracheostomy, ventilator use, non-invasive mechanical ventilator use (BiPAP, CPAP, Airvo), diaphragmatic pacing, oxygen

Exclusion Criteria:

* Other caretakers such as grandparents, aunts, uncles

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Parents of technology dependent pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of pediatric patient getting COVID 19 vaccine | 6 months after initial survey

SECONDARY OUTCOMES:
Percentage of mothers getting COVID 19 vaccine | 6 months after initial survey
Percentage of fathers getting COVID 19 vaccine | 6 months after initial survey
Percentage of other adults in household getting COVID 19 vaccine | 6 months after initial survey
Percentage of other eligible children in household getting COVID 19 vaccine | 6 months after initial survey

CONTACTS AND LOCATIONS:
Overall Officials: Karen Capusan, MSN, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Physician Partners, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dosanjh A. Pediatric Vaccine Hesitancy and the Utilization of Antibody Measurements: A Novel Strategy with Implications for COVID 19. J Asthma Allergy. 2021 Apr 23;14:427-431. doi: 10.2147/JAA.S303309. eCollection 2021. PMID 33935504
- [Background] Khubchandani J, Sharma S, Price JH, Wiblishauser MJ, Sharma M, Webb FJ. COVID-19 Vaccination Hesitancy in the United States: A Rapid National Assessment. J Community Health. 2021 Apr;46(2):270-277. doi: 10.1007/s10900-020-00958-x. Epub 2021 Jan 3. PMID 33389421
- [Background] McAteer J, Yildirim I, Chahroudi A. The VACCINES Act: Deciphering Vaccine Hesitancy in the Time of COVID-19. Clin Infect Dis. 2020 Jul 28;71(15):703-705. doi: 10.1093/cid/ciaa433. PMID 32282038
- [Background] Vasconcello-Castillo L, Torres-Castro R, Vera-Uribe R, Paiva R. COVID-19: Precautions with children in home mechanical ventilation. Pediatr Res. 2020 Oct;88(4):520-521. doi: 10.1038/s41390-020-1047-7. Epub 2020 Jul 2. No abstract available. PMID 32615580